CLINICAL TRIAL: NCT01038232
Title: Measuring Distress Tolerance With Functional MRI
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Maryland, College Park (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910453; 10-DA-N453
Record Dates: First submitted 2009-12-19; First posted 2009-12-23 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2015-03-24

CONDITIONS: Cocaine Dependence
Keywords: Distress Tolerance; Cocaine Dependence; Relapse; Limbic System; Prefrontal Cortex; Healthy Volunteer; HV
MeSH Terms: conditions — Cocaine-Related Disorders; Recurrence

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- People who are in treatment for substance abuse often feel distress during the withdrawal period and afterward. Some individuals feel distress more acutely than others, and this distress has been linked to poor treatment outcomes and increased risk of relapse in smokers, alcoholics, and cocaine- and heroin-dependent individuals. More research is needed on the effects of distress on the brain, particularly in individuals who are seeking treatment for substance abuse. Researchers are interested in using functional magnetic resonance imaging (fMRI) scanning to study distress tolerance in both substance users seeking treatment and healthy non-drug-using volunteers.

Objectives:

- To use functional magnetic resonance imaging to study the effectiveness of a distress tolerance assessment.

Eligibility:

- Individuals between 18 and 50 years of age who are either cocaine dependent or healthy non-drug-using volunteers.

Design:

* This study involves an initial screening visit and a scanning visit, with four followup visits.
* Participants will be screened with a medical history and physical examination, as well as blood samples and questionnaires about mood and past and current drug use.
* Participants will have a structural MRI scan of the brain to provide a baseline reading for comparison. Participants will then have an fMRI scanning session, which will include both the distress tolerance assessment and relevant control tasks. Heart rate, blood pressure, and other physical reactions will be monitored throughout the scan. Participants will also provide blood and saliva samples to measure stress hormone levels.
* Participants will be eligible to have followup assessments with fMRI scanning 1, 3, 6, and 12 months after the scanning visit.

DETAILED DESCRIPTION:
Objective: The primary objective of the current study is to implement a distress tolerance assessment for use in fMRI to determine the neurobiological differences between individuals with low and high distress tolerance. Additionally, other biological and physiological indicators will be assessed, including genetic polymorphisms, salivary cortisol, galvanic skin response, and blood pressure. The overall hypothesis is that individuals with low distress tolerance will exhibit hyperactivation in the extended amygdala and hypoactivation of the prefrontal cortex and anterior cingulate cortex when experiencing affective distress and failure during a stressful task, as compared to individuals with high distress tolerance.

Study Population: The study population will consist of healthy male and female adult volunteers (18-55 years old), as well as an otherwise healthy sample of male and female treatment seeking substance users with cocaine users (18-55 years old) (see exclusion criteria).

Experimental Design and Methods: After being medically cleared and giving written informed consent, each participant will undergo a structural MRI scan of the brain, and undergo an fMRI scanning session, which will include administration of the distress tolerance and relevant control tasks. Physiological response to the tasks, including heart rate, blood pressure, galvanic skin conductance, and salivary cortisol concentrations will be monitored throughout the fMRI scan. Follow-up assessments on control and cocaine dependent participants will occur at 1, 3, 6, and 12 months after the baseline assessment. Genetic data collected under the aegis of protocol 10-DA-N457 will be compared with data collected under this study.

Outcome Measures: Outcome measures include distress tolerance measured as latency in seconds to task termination on each of the distress tolerance tasks, neural indices of distress tolerance (for all participants), and substance use treatment outcomes (for cocaine users) including relapse to drug use, latency to first cocaine use, and number of substance use days per week at follow-ups.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Be between the ages of 18 and 55.
  2. Be in good health.
  3. Be right-handed.
  4. Cocaine dependent participants: Endorse regular cocaine use (i.e., greater than or equal to 2 times per week) in the past year.
  5. Non-drug using controls: will be matched to the cocaine using participants with respect to age, gender, IQ, socioeconomic factors, and years of education.

EXCLUSION CRITERIA:

1. Pregnant. Urine pregnancy tests will be performed on all female volunteers of child-bearing age before each experimental session.
2. Have implanted metallic devices (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted metal parts) or claustrophobia rendering them unable to undergo fMRI scanning.
3. Have major medical illnesses to include, but not limited to, hypertension, cardiovascular disease, asthma, diabetes, peripheral vascular diseases, coagulopathies, syncope, history of superficial or deep vein thrombosis, HIV, or other clinically significant infectious diseases.
4. Have current major psychiatric disorders to include, but not limited to, mood, anxiety, borderline personality disorder, psychotic disorders, or substance-induced psychiatric disorders,
5. Have neurological illnesses including, but not limited to, seizure disorders, migraine, multiple sclerosis, movement disorders, or history of head trauma, CVA, CNS tumor.
6. Control participants: Meet DSM-IV criteria for any past or current substance abuse or dependence; use of illicit substances in the last 30 days or nicotine if use is greater than 10 cigarettes per day and/or Fagerstrom score is greater than 3.
7. Cocaine using participants:

   1. Non-treatment subjects: Meet DSM-IV criteria for substance dependence on any substance other than nicotine or cocaine in the month prior to study enrollment. Only (except nicotine or cocaine dependence will be allowed in the month prior to enrollment. Current abuse on any substance will be acceptable.). While it might be preferable to exclude individuals whose use of other substances reaches the threshold of abuse, inclusion of such individuals will not necessarily contaminate the data.
   2. Inpatient cocaine subjects: Those who meet DSM-IV TR criteria for the course specifier In a Controlled Environment may have a history of dependence on substances other than cocaine before their admission to the inpatient treatment program.
8. Regular use of any prescription, over-the-counter, or herbal medication that may alter CNS function, cardiovascular function or neuronal-vascular coupling. Medications that could interfere with the BOLD signal include compounds that have been shown to be vasoactive, including alpha agonists, beta blockers, and calcium channel blockers.
9. Have cognitive impairment as assessed by screening WASI vocabulary subtest below 48, corresponding to full IQ of 85 (in that case on screening, a full WASI will be done to verify IQ of 85 or above).
10. Acute drug intoxication or positive urine drug screen at the beginning of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2009-12-04; Study Completion 2015-03-24

PRIMARY OUTCOMES:
To identify neural indices of distress tolerance using fMRI in healthy non-drug users, and examine the relationship between these neural indices and important physiological, biological, and behavioral correlates of distress tolerance.

SECONDARY OUTCOMES:
To determine if neural processes associated with distress tolerance predict sustained abstinence among treatment seeking cocaine dependent participants following 1, 3, 6, and 12 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (2):
- United States (2):
  - National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland
  - University of Maryland, College Park, College Park, Maryland

REFERENCES:
- [Background] Abercrombie HC, Schaefer SM, Larson CL, Oakes TR, Lindgren KA, Holden JE, Perlman SB, Turski PA, Krahn DD, Benca RM, Davidson RJ. Metabolic rate in the right amygdala predicts negative affect in depressed patients. Neuroreport. 1998 Oct 5;9(14):3301-7. doi: 10.1097/00001756-199810050-00028. PMID 9831467
- [Background] Ahmed SH, Koob GF. Cocaine- but not food-seeking behavior is reinstated by stress after extinction. Psychopharmacology (Berl). 1997 Aug;132(3):289-95. doi: 10.1007/s002130050347. PMID 9292629
- [Background] Acker C. Neuropsychological deficits in alcoholics: the relative contributions of gender and drinking history. Br J Addict. 1986 Jun;81(3):395-403. doi: 10.1111/j.1360-0443.1986.tb00346.x. No abstract available. PMID 3461848